CLINICAL TRIAL: NCT06043505
Title: Impact of an Echographic Algorithm on Hemodynamic Optimization in the First 4 Days of Septic Shock Management: a Multicentric, Randomized, Controlled, Open Label Pilot-study
Brief Title: Impact of an Echographic Algorithm on Hemodynamic Optimization in the First 4 Days of Septic Shock Management
Acronym: STOPFLUID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-A00111-44
Record Dates: First submitted 2023-06-30; First posted 2023-09-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Shock, Septic; Hemodynamic Instability
Keywords: Monitoring; Transthoracic Echocardiography; Blood Volume; Fluid management
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Strategy: STOPFLUID Algorithm (Experimental): Fluid management is optimised using the specific echographic hemodynamic algorithm ('STOPFLUID') of this study described during the first 4 days of septic shock. Fluid bolus will not be administered in case of increased left ventricle filling pressures; fluid challenge will be performed based on dynamic indices and fluid depletion will be considered on the basis of Lung UltraSound (LUS) assessment.
  Interventions: Other: Echographic hemodynamic algorithm guiding fluid resuscitation
- Standard Strategy (No Intervention): Fluid management will be handled according to standard care, without using transthoracic echocardiography (TTE) during the first 4 days of septic shock management. Haemodynamic monitoring including pulmonary artery catheter, transpulmonary thermodilution, or any other device will be left at the physician's discretion. TTE will be allowed in the standard group only for excluding cardiac tamponade in case of clinical suspicion (one or more of the following signs: jugular distension, pulsus paradoxus)

INTERVENTIONS:
Other: Echographic hemodynamic algorithm guiding fluid resuscitation — Ultrasound Hemodynamic Algorithm (UHA):
  1. st step: 1/ Assessment of left ventricular filling pressures by Mitral Doppler echocardiography (2) 2/ Pulmonary ultrasound on 4 anterior dials (3)
     E/Ea >14 and/or E/A >2
     * YES => No filling test => Bilateral anterior B lines on lung ultrasound => YES => Consider administration of diuretics
     * NO => Step 2
  2. nd step: Assessment of filling response by dynamic maneuvers VTI (Velocity Time Integral) increase >15% after passive leg raising (4) or Mini-fluid challenge (5,6) Or decision of a 250ml filling test
     * YES => consider 250ml bolus filling
     * NO => stop vascular filling
  3. rd step if dynamic maneuvers in favor of a response to filling: 1/ Assessment of response to 250ml filling 2/ If no response to vascular filling: Pulmonary ultrasound on 4 anterior dials (3) Change from a pulmonary profile A to a pulmonary profile B
     * YES => depletion
     * NO => stop vascular filling
  Arms: Interventional Strategy: STOPFLUID Algorithm

SUMMARY:
Fluid management is one of the key issues in the initial management of septic shock (SS). Fluid overload and hypovolemia have been associated with increased mortality in several trials. Transthoracic echocardiography (TTE) and lung ultrasound are recommended for haemodynamic assessment in critically ill patients. However, the benefit of hemodynamic optimisation using echography has not been yet evaluated. The purpose of this multicenter, controlled, randomized trial is to assess the impact of an echocardiographic algorithm of hemodynamic optimization on fluid management in septic patients during the first 4 days of therapy.

ELIGIBILITY:
All eligible patients will have a cardiac echocardiogram prior to inclusion for the sole purpose of eliminating special situations that are part of the non-inclusion criteria listed below.

Inclusion Criteria

* Patient in an intensive care unit who develops septic shock on admission or during hospitalization, as defined by SEPSIS-3 criteria.
* Patient or trusted person / legal representative / family member / curator / guardian who has given free and informed consent and has signed the consent form or patient included in an emergency situation.
* Patient affiliated or beneficiary of a health insurance plan.
* Patient at least (≥) 18 years of age.

Exclusion Criteria:

* Refusal of consent.
* Patient under court protection or guardianship.
* Moribund patient with a life expectancy of less than 48 hours.
* Non-echogenic patient.
* Cardiac tamponade.
* Infective endocarditis.
* Intracavitary thrombus.
* Dilated cardiomyopathy with LVEF (Left Ventricular Ejection Fraction<40%.
* Parturient or nursing patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-10-26 (Estimated)

PRIMARY OUTCOMES:
Volume of vascular filling during the first 4 days | Day 4
  This takes into account the cumulative volume of vascular filling administered to improve cardiac output during the 4 first days, measured in Liter (L)

SECONDARY OUTCOMES:
.Analysis of the primary endpoint related to ARDS ([acute respiratory distress syndrome, according to Berlin criteria) | Day 4
  Analysis of the primary endpoint in relation with presence or absence of ARDS at inclusion
Analysis of the primary endpoint related to severe renal dysfunction | Day 4
  Analysis of the primary endpoint in relation with severe renal dysfunction defined as a KDIGO (Kidney Disease Improving Global Outcomes) score ≥3 vs <3.
Analysis of the primary endpoint in relation with patient severity | Day 4
  Analysis of the primary endpoint in relation withpatient severity according to SAPS 2 (Simplified Acute Physiology Score) score: <15, 15-30, >30
Mortality | Day 28
  Patient deceased: yes or no
Number of days alive without failure at Day 28 | Day 28
  Number of days without failure
Time to normalization of lactatemia (<2 mmol/l) | Day 4
  Represents time from randomization to first lactatemia <2 mmol/l in hours
Fluid balance in L | Day 4
  The fluid balance will be deduced from the daily weight changes in kilograms, the density of water being equal to 1
Therapeutic adjustments including bolus vascular filling, changes in vasopressor flow, and administration of diuretics | Day 4
  Number of therapeutic adjustments
Length of stay in ICU (ready for discharge) | Day 28
  Length of stay in ICU from randomization to discharge in days
Length of stay in hospital | Day 28
  Number
Adverse effects | Day 28
  Number and type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, Madsen KR, Moller MH, Elkjaer JM, Poulsen LM, Bendtsen A, Winding R, Steensen M, Berezowicz P, Soe-Jensen P, Bestle M, Strand K, Wiis J, White JO, Thornberg KJ, Quist L, Nielsen J, Andersen LH, Holst LB, Thormar K, Kjaeldgaard AL, Fabritius ML, Mondrup F, Pott FC, Moller TP, Winkel P, Wetterslev J; 6S Trial Group; Scandinavian Critical Care Trials Group. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. N Engl J Med. 2012 Jul 12;367(2):124-34. doi: 10.1056/NEJMoa1204242. Epub 2012 Jun 27. PMID 22738085
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Douglas IS, Alapat PM, Corl KA, Exline MC, Forni LG, Holder AL, Kaufman DA, Khan A, Levy MM, Martin GS, Sahatjian JA, Seeley E, Self WH, Weingarten JA, Williams M, Hansell DM. Fluid Response Evaluation in Sepsis Hypotension and Shock: A Randomized Clinical Trial. Chest. 2020 Oct;158(4):1431-1445. doi: 10.1016/j.chest.2020.04.025. Epub 2020 Apr 27. PMID 32353418
- [Background] Muller L, Toumi M, Bousquet PJ, Riu-Poulenc B, Louart G, Candela D, Zoric L, Suehs C, de La Coussaye JE, Molinari N, Lefrant JY; AzuRea Group. An increase in aortic blood flow after an infusion of 100 ml colloid over 1 minute can predict fluid responsiveness: the mini-fluid challenge study. Anesthesiology. 2011 Sep;115(3):541-7. doi: 10.1097/ALN.0b013e318229a500. PMID 21792056
- [Background] Biais M, de Courson H, Lanchon R, Pereira B, Bardonneau G, Griton M, Sesay M, Nouette-Gaulain K. Mini-fluid Challenge of 100 ml of Crystalloid Predicts Fluid Responsiveness in the Operating Room. Anesthesiology. 2017 Sep;127(3):450-456. doi: 10.1097/ALN.0000000000001753. PMID 28640019
- [Background] Lichtenstein DA, Meziere GA, Lagoueyte JF, Biderman P, Goldstein I, Gepner A. A-lines and B-lines: lung ultrasound as a bedside tool for predicting pulmonary artery occlusion pressure in the critically ill. Chest. 2009 Oct;136(4):1014-1020. doi: 10.1378/chest.09-0001. PMID 19809049